CLINICAL TRIAL: NCT01911884
Title: Assessment of Quality of Global and Sexual Life and Impact of Surgical and Non Surgical Vaginal Aplasia in Patients With a Rokitansky Syndrome
Acronym: MRKH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P110124; ID RCB : 2011-A01517-34
Record Dates: First submitted 2013-07-26; First posted 2013-07-30 (Estimated); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Rokitansky Syndrome; Surgical or Vaginal Dilatation of Vaginal Aplasia
Keywords: Rokitansky syndrome; surgical or vaginal dilatation of vaginal aplasia; quality of global and sexual life
MeSH Terms: conditions — Mullerian aplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with a Rokitansky Syndrome (Other): Patients with a Rokitansky Syndrome
  Interventions: Behavioral: evaluate quality of life of surgical and non surgical vaginal aplasia

INTERVENTIONS:
Behavioral: evaluate quality of life of surgical and non surgical vaginal aplasia — protocol designed to evaluate quality of life of surgical and non surgical vaginal aplasia

SUMMARY:
The principal objective is to assess the general health status and the sexual health status of women with Rokitansky syndrome having received a surgical or non surgical treatment.

The secondary purpose is to assess the anatomical aspect and the quality of sexual life. To search a correlation between the anatomical result, the general and sexual quality of life. To compare the different techniques of medical follow-up in terms of anatomic results, general quality of life, sexual quality of life, complications and morbidities.

To evaluate social inclusion of these women with their family situation, social and professional category and their job.

At the same time, we propose an evaluation with a psychologist to study the impact of the announcement of the diagnosis. This impact study is conducted at a distance from diagnosis.

DETAILED DESCRIPTION:
The MRKH syndrome is a congenital disorder characterized by absence of uterus and at least the two thirds of the vagina, a female phenotype and a normal karyotype XX.

These patients have normal ovaries and fallopian tubes. The external genitalia are normal. This syndrome was described by Mayer (1829), Rokitansky ( 1838), Kuster ( 1910) and Hauser ( 1961). About one in every 4500 female babies has this condition. This syndrome represents 85% of congenital vagina aplasia and is the second cause of primary amenorrhea after disorders of sexual development. These women are unfertile.

The malformation can be isolated or associated with other malformations called MURCS (Müllerian duct aplasia, renal aplasia, and cervicothoracic somite dysplasia), as kidney ( 30%), bone ( 10%) or cardiac malformations ( 1%).

The most common age for MRKH to be diagnosed is when the woman hasn't started her period ( 85%).Some girls may find out at an earlier age when there is a severe malformation , during a systematic gynaecological examination or during an pelvic ultrasound. When the women are older, the syndrome can be diagnosed during studies for infertility.

A pelvic ultrasound is usually the first test performed to assess presence of uterus. A magnetic resonance imaging may be used to complete the investigations. These tests can also confirm if there are two ovaries and two kidneys. Sometimes, a very small uterus can be seen, it's a uterine horn.

The psychological management is essential to take care of the women affected.It seeks to understand the impact of the diagnosis announcement and the various treatments offered. The follow-up can be different for each girl and her parents during several appointments.

Therapeutic management can be proposed when the girl is ready because the therapeutic is long and difficult. Two therapeutic approaches can be proposed: to create a vagina using dilators or having a surgical procedure. In France, vaginal reconstruction with dilators is the most used. This method consists in dilating the vagina progressively with different sizes of dilators in order to obtain a vaginal opening of 8 cm around 6 months after treatment initiation. This method is successful in about 75% of cases. Complications are exceptional.

Surgery is an option for patients who are unsuccessful with dilatators or patients who prefer surgery. A number of operations are appropriate for the correction of vaginal agenesis. Vecchietti procedure and sigmoid vaginoplasty are the most commonly used techniques in France.

In national and international publications, it is impossible to compare scientifically the results of the different technique because of the small effective in each studies and because of the the lack of standardized assessment. Studies report the functional result for each technique but none compare the techniques used. No studies compared the result in terms of anatomical and function results, complications and quality of life.

The demonstration of a positive correlation between the anatomic criteria and the functional results would help to guide the surgical technique. The lack of correlation would suggest that a perfect anatomical reconstruction is not essential. If it is demonstrated, the management should focus on other criteria like psychological management. Several factors seem to influence the general and sexual quality of life of women affected by the Rokitansky syndrome. Our objective is to evaluate the importance of these factors to improve the treatment of these women.

ELIGIBILITY:
Inclusion Criteria:

* Patient affected with Rokitansky syndrome
* Patient over 18 years old
* Patient care with dilatations or by surgery since 1995
* Patient having started dilatations or having had surgery since at least one year
* Patient who signed the consent
* French patient
* Women with social welfare

Exclusion Criteria:

* Patient with a serious chronic disease interfering with analysis to be performed in this project.
* Patient can't reading or writing
* Patient with legal protection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2012-10-11 (Actual); Primary Completion 2015-04-10 (Actual); Study Completion 2015-04-10 (Actual)

PRIMARY OUTCOMES:
Assessment of quality of global life | Day 0
  To fill a self-administered questionnaire: the World Health Organization Quality Of Life (general scale WHOQOL)

SECONDARY OUTCOMES:
Assessment of quality of sexual life | Day 0
  To fill 2 self-administered questionnaires : Female Sexual Function Index and Female Sexual Dysfunction Scale-Revised (FSFI and FSDS)
Assessment of anatomic results | Day 0
  Gynaecological examination
Assessment of social integration | Day 0
  To fill a self-administered questionnaire (marital status, occupational group, education level, employment status)

CONTACTS AND LOCATIONS:
Overall Officials: Michel POLAK, PUPH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service d'Endocrinologie et Gynécologie Pédiatriques Hôpital Necker Enfants Malades, Paris, France

REFERENCES:
- [Background] Cheikhelard A, Bidet M, Baptiste A, Viaud M, Fagot C, Khen-Dunlop N, Louis-Sylvestre C, Sarnacki S, Touraine P, Elie C, Aigrain Y, Polak M; French MRKH Study Group. Surgery is not superior to dilation for the management of vaginal agenesis in Mayer-Rokitansky-Kuster-Hauser syndrome: a multicenter comparative observational study in 131 patients. Am J Obstet Gynecol. 2018 Sep;219(3):281.e1-281.e9. doi: 10.1016/j.ajog.2018.07.015. Epub 2018 Jul 21. PMID 30036500